CLINICAL TRIAL: NCT04942171
Title: EMOTIon and COgNitive Function After Atrial Fibrillation Catheter Ablation vs. Medical Therapy; Randomized Clinical Trial (EMOTICON Trial)
Brief Title: EMOTIon and COgNitive Function After Atrial Fibrillation Catheter Ablation vs. Medical Therapy(EMOTICON Trial)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-1488
Record Dates: First submitted 2021-05-26; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atrial fibrillation catheter ablation group (Experimental): catheter ablation
  Interventions: Procedure: Atrial fibrillation catheter ablation group
- Medical therapy group (Active Comparator): standard treatment include anti-arrhythmic drug
  Interventions: Drug: Medical therapy group

INTERVENTIONS:
Procedure: Atrial fibrillation catheter ablation group — 1. Pulmonary vein isolation
  2. Additional treatment for lesions caused by non-pulmonary veins
  3. Esophageal temperature monitoring to prevent damage to the esophagus
  4. Evaluation of procedure time and radiofrequency ablation time
  5. Evaluation of complications after the procedure
  6. Rhythm follow-up after the procedure is conducted in accordance with the above study design.
  7. Conduct a survey on cognitive function and emotion before and 12 months after the procedure
  Arms: Atrial fibrillation catheter ablation group
Drug: Medical therapy group — 1. Use of beta-blockers or calcium channel blockers for pulse rate control
  2. Antiarrhythmic drugs are administered to patients with highly symptomatic atrial fibrillation symptoms even after pulse rate control.
  3. If symptoms are not controlled even with antiarrhythmic drugs, electrical conversion to restore sinus rhythm.
  4. To prevent cerebral infarction, maintain optimal anticoagulant therapy according to the risk score for cerebral infarction.
  5. Conduct a questionnaire on cognitive function and emotion before and 12 months after the procedure
  Arms: Medical therapy group

SUMMARY:
"Atrial fibrillation (AF) is an arrhythmic disease that increases especially in the elderly, increasing the risk of ischemic stroke by 5 times and is a major cause of dementia and cognitive impairment.

Cognitive dysfunction accompanying AF occurs regardless of the presence or absence of stroke, and AF itself is known to affect cognitive function.

However, since cognitive dysfunction is also affected by various accompanying chronic diseases, whether the cognitive dysfunction accompanying AF is due to subclinical ischemic stroke, cerebral hypoperfusion due to reduced cardiac output, inflammatory reaction or platelet dysfunction are unclear.

Recently, this research team reported an improvement in cognitive function with active sinus rhythm therapy such as AF catheter ablation. Nevertheless, it has not yet been proven whether such active and invasive AF treatment affects the improvement of cognitive function or depression by a randomized clinical trial.

In this prospective randomized clinical comparative study, the investigators will compare the AF catheter ablation group and drug therapy group in terms of cognitive function tests and depression psychological tests at baseline and a year after treatment. Our hypothesis is that AF catheter ablation is superior to drug therapy to improve cognitive function and depressive mood.

DETAILED DESCRIPTION:
Study design

1. Prospective randomization (catheter ablation group vs. drug treatment group) (Python program is used, the random number module is imported using the import random syntax, and the random number table of the two groups is prepared and used)
2. Target number of targets 320 (160 for each group)
3. Cardiac rhythm follow-up: 2012 ACC/AHA/ESC guidelines (baseline, 3 months, every 6 months after Holter, Electrocardiogram when symptoms are present)
4. Anticoagulant therapy follows 2014 ACC/AHA/ESC guidelines.
5. Evaluation of MOCA score (cognitive function), CES-D score (depression), and GAD-7 score (anxiety) at baseline and a year after treatment, respectively.
6. Evaluation of all adverse events occurring in each group, hospitalization rate, major cardiovascular attack, and mortality rate comparison

Progress and rhythm/ ECG follow-up

1. Implemented in accordance with 2012 ACC/AHA/HRS guidelines for AF management
2. Baseline MOCA, CES-D, and GAD-7 score evaluation
3. Outpatient follow-up observation 1 to 2 weeks after the start of the procedure or medication
4. Follow-up observation at intervals of 2 months, 6 months, and then every 6 months after starting the procedure or medication
5. If the patient complains of arrhythmia symptoms, conduct an electrocardiogram at any time, and follow the rhythm with a Holter or event recorder.
6. Follow-up MOCA, CES-D, and GAD-7 score evaluation

Follow-up observation

* All patients are scheduled to visit the outpatient clinic every 6 months after 1~2 weeks, 2 months, 6 months, and even if they have symptoms in the middle, they will be treated as an outpatient at any time.
* An ECG is administered at every outpatient visit. A 24-hour Holter or event recorder was administered for 1 year at intervals of 2, 6, and 6 months after the procedure (2012 Heart Rhythm Society/EHRA/European Cardiac Arrhythmia Society Expert Consensus Statement guidelines).
* If atrial fibrillation or atrial tachycardia lasting more than 30 seconds is observed on a standard electrocardiogram, event electrocardiogram, or Holter, it is evaluated as recurrence. Recurrence within 3 months after the procedure is classified as early recurrence, and recurrence after 3 months is classified as clinical recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 20 and 80 years of age who have appropriate indication for catheter ablation for AF
2. AF patients with left atrium diameter <55 mm
3. Antiarrhythmic drug-resistant AF
4. Anticoagulation eligible patients

Exclusion Criteria:

1. AF associated with severe cardiac malformation or structural heart disease
2. Patients undergoing treatment for cognitive disorders, emotional disorders, and anxiety disorders
3. Patients with severe renal dysfunction or difficulty in CT imaging using contrast media
4. Patients with a previous history of AF ablation or other open heart surgery
5. Patients with active internal bleeding
6. Anticoagulant therapy not eligible patients
7. Valvular AF (mitral valve stenosis>grade 2, mechanical valve, mitral valve reconstruction)
8. Significant comorbidities
9. Patients with an expected survival period of less than 1 year
10. Drug or alcohol addiction patients
11. Among eligible persons, those who cannot read the consent form (illiteracy, foreigners, etc.)
12. Patients judged to be unsuitable for participation in clinical research based on the judgment of other researchers

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive function, depression, and anxiety scale after catheter ablation or drug treatment after 1 year of randomization | 1 year
  Compasison of scale change using the Moca questionnaire.
Changes in depression scale after catheter ablation or drug treatment after 1 year of randomization | 1 year
  Compasison of scale change using the CES-D questionnaire.
Changes in anxiety scale after catheter ablation or drug treatment after 1 year of randomization | 1 year
  Compasison of scale change using the GAD-7 questionnaire.

SECONDARY OUTCOMES:
Differences according to AF type | 1year
Differences in adverse effects of ablation vs. medications | 1year
Differences in MACE, Death, and Readmission rate | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Nam Pak, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided